CLINICAL TRIAL: NCT04431570
Title: Repetitive Transcranial Magnetic Stimulation for the Treatment of Freezing of Gait in Parkinson's Disease: A Randomized Controlled Trial
Brief Title: Repetitive Transcranial Magnetic Stimulation for the Treatment of Freezing of Gait in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: rTMSPDFOG-PUMCH
Record Dates: First submitted 2020-04-27; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Parkinson Disease; Gait Disorders, Neurologic
Keywords: freezing of gait; FMRI; rTMS
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- rTMS over M1 region (Experimental): The stimulus intensity was set to 100% of the resting motor threshold. Ten sessions of rTMS were delivered over 2 weeks, one session per day for 5 consecutive days per week. Each session consisted of 10 trains of 100 pulses at 10Hz with an inter-train interval of 40 seconds. In this group, the target of rTMS is M1 region.
  Interventions: Device: rTMS
- rTMS over supplementary motor area (SMA) (Experimental): The stimulus intensity was set to 100% of the resting motor threshold. Ten sessions of rTMS were delivered over 2 weeks, one session per day for 5 consecutive days per week. Each session consisted of 10 trains of 100 pulses at 10Hz with an inter-train interval of 40 seconds. In this group, the target of rTMS is SMA region.
  Interventions: Device: rTMS
- sham stimulation (Sham Comparator)
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: rTMS — The device is made in London, United Kingdom
  Arms: rTMS over M1 region; rTMS over supplementary motor area (SMA)
Device: sham stimulation — the device of sham stimulation was MagStim MC-P-B70 placebo butterfly coil
  Arms: sham stimulation

SUMMARY:
Freezing of gait (FOG) is a common and devastating symptom in advanced stage Parkinson's disease (PD), which contributes to falls and disability. Unfortunately, there is no effective pharmacological treatment for FOG. It is suggested that the cortex-basal ganglia circuit, especially the frontal lobe, plays an important role in the pathogenesis of FOG. Repetitive transcranial magnetic stimulation (rTMS) effects over the cortex and affects the subcortical neural circuits. Previous studies have demonstrated that rTMS can improve FOG for PD patients. In the present randomized controlled trial (RCT) study, the invastigators aim to investigate the efficiency of rTMS over different motor regions of frontal lobe. The efficacy of treatment is evaluated by the score of FOG questionnaire and FOG provoking test, and the changing of neural network shown by functional magnetic resonance imaging (FMRI). Then the effects of rTMS over different brain regions will be compared for choosing a better target. The study will provide the evidence for non-invasive neuro-modulation of Parkinson's disease with freezing of gait (PD-FOG).

ELIGIBILITY:
Inclusion Criteria:

* Subjects fulfilled the diagnosis of idiopathic Parkinson's disease according to MDS-PD criteria
* Hoehn & Yahr (H-Y) stage was 2 or 3
* All subjects had freezing of gait which was identified by FOGQ

Exclusion Criteria:

* cognitive impairment (MMSE score<22) or major depression (HAMD-24 score>25)
* severe visual and/or haring impairment
* significant medical or psychiatric illnesses
* history of deep brain stimulation (DBS) surgery or pacemaker implantation. MRI cannot be performed in those patients
* current treatment with medication cannot be maintained during the study

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-06-15 (Estimated); Primary Completion 2022-04-14 (Estimated); Study Completion 2022-06-14 (Estimated)

PRIMARY OUTCOMES:
the change of freezing of gait questionnaire (FOGQ) | through study completion, an average of 2 weeks
  a self-assessment scale for evaluating FOG severity，the minimum value is 0, the maximum value is 24, and higher scores mean a worse outcome.

SECONDARY OUTCOMES:
the change of freezing of gait score (FOG score) | through study completion, an average of 2 weeks
  assess the severity of FOG, the minimum value is 0, the maximum value is 36, and higher scores mean a worse outcome.
the change of score of Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III | through study completion, an average of 2 weeks
  assess the motor ability, the minimum value is 0, the maximum value is 132, and higher scores mean a worse outcome.
the change of Hamilton Depression (HAMD) Scale | through study completion, an average of 2 weeks
  assess the severity of depression, the minimum value is 0, the maximum value is 76, and higher scores mean a worse outcome.
the change of Mini-mental State Examination (MMSE) scale | through study completion, an average of 2 weeks
  assess the severity of mental state, the minimum value is 0, the maximum value is 30, and higher scores mean a worse outcome.
the change of Parkinson's Disease Questionnaire (PDQ-39) | through study completion, an average of 2 weeks
  assess the quality of life, the minimum value is 0, the maximum value is 156, and higher scores mean a worse outcome.
functional image of the brain (FMRI) | through study completion, an average of 10 days
  graph theoretical analysis of the brain network

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China